CLINICAL TRIAL: NCT06789523
Title: Friendship Bench for Women Who Use Methamphetamine in Vietnam
Acronym: FB-WWUM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hanoi Medical University (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH); University of North Carolina, Chapel Hill (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K43TW012620-01A1 (NIH); K43TW012620-01A1 (NIH)
Record Dates: First submitted 2024-12-12; First posted 2025-01-23 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Methamphetamine Use; Common Mental Disorders (CMD)
Keywords: methamphetamine; women who use drugs; common mental disorders; Friendship Bench; lay worker-delivered intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Friendship Bench (Experimental): Participants randomized to the intervention condition will receive the adapted Friendship Bench intervention.
  Interventions: Behavioral: Friendship Bench
- Usual psychiatric care (Active Comparator): Participants in the control group will receive usual care for their common mental disorders.
  Interventions: Behavioral: Usual psychiatric care

INTERVENTIONS:
Behavioral: Friendship Bench — The Friendship Bench model comprises 6 weekly, individual sessions with trained peer workers in addition to the usual care. Peer workers will help participants identify problems, outline potential solutions, and implement selected solutions.
  The adaptation of Friendship Bench for Vietnamese methadone patients made revisions, such as removing the 'Belief in supernatural powers' section, replacing the Shona Symptom Questionnaire with DASS-21, and adding meth use. But this adaptation removed women-focused content on pregnancy and postpartum depression that we plan to include.
  Arms: Friendship Bench
Behavioral: Usual psychiatric care — Usual care includes monthly check-ups by peer workers, referral to hospital-based psychiatric services or other available mental health services if needed. This usual care might surpass standard psychiatric care in other provinces given that peer workers in Haiphong have been well trained on case management skills.
  Arms: Usual psychiatric care

SUMMARY:
The high comorbidity of mental health issues and meth use in women worsens both their mental health and meth use outcomes. The study team proposes to evaluate the potential of Friendship Bench to be used as a low-threshold, task-shifting mental health intervention among women who use methamphetamine in Vietnam - a lower-middle-income country. The study will provide preliminary data for a R01 trial testing the effectiveness Friendship Bench to improve mental health and methamphetamine use outcomes among women who use methamphetamine in Vietnam.

DETAILED DESCRIPTION:
The specific aims of this research proposal are to: (1) assess the mental health needs of WWUM in Haiphong, (2) adapt Friendship Bench to the specific needs of Vietnamese WWUM and (3) assess the feasibility, fidelity, and acceptability of the adapted Friendship Bench for common mental disorders among WWUM and preliminary indicators of its impact in improving their mental health and methamphetamine use in a two-arm randomized trial, comparing Friendship Bench with usual psychiatric care.

ELIGIBILITY:
Inclusion Criteria:

* Adult women (>=18 years old)
* Moderate or greater risk for meth use (ASSIST ≥ 4)
* Moderate or greater CMD symptom severity (Depression ≥ 10, Anxiety ≥ 8, and/or Stress ≥ 15 on DASS-21)

Exclusion Criteria:

* Severe psychotic disorders or other interfering problems that require specialty care;
* Inability to understand study procedures by the research team's judgment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study focuses on women who use methamphetamine.
Enrollment: 100 (Estimated)
Dates: Start 2025-06-11 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility: the ability to enroll women who use meth with common mental disorders in the pilot | From enrollment to the end of intervention at 6 weeks
  The ability to enroll WWUM is assessed through the recruitment rate (number of WWUM approached to accrue the final sample) and reasons for non-participation.
Feasibility: the ability to retain WWUM with common mental disorders in the pilot | From enrollment to the end of intervention at 6 weeks
  Based on data from previous studies in Vietnam, the study team defines feasible retention as 80% retention at 6-weeks.
Feasibility: adequate completion of Friendship Bench sessions | From enrollment to the end of intervention at 6 weeks
  As peer outreach workers will conduct home visits or visits to workplace, the study team considers 70% participants attending all 6 individual sessions to be feasible. The reasons for session non-attendance, and counselor time per session and per patient including preparation, documentation, and supervision will also be assessed to explain the Friendship Bench completion rate.
Acceptability | At Week 6
  Acceptability is defined as the perception among implementation stakeholders that the intervention is agreeable or satisfactory. The study team will assess acceptability through the 6-week follow-up interview with all participants (n=100) and peer workers (n=10). Acceptability will also be assessed qualitatively using the post-intervention in-depth interviews with peer workers (n=10), participants (n=20) and brief exit interviews with supervisors (n=2). The interviews will assess how easy the intervention is to participate and to deliver, the perceived usefulness of the intervention and suggestions for improvement. Intervention acceptability is defined as 80% participants rating the intervention as acceptable and by a common theme of positive perceptions of Friendship Bench in qualitative data.
Fidelity | From enrollment to the end of intervention at 6 weeks
  Fidelity is defined as delivery of the intervention as intended. Master trainers will use a checklist to assess fidelity to session content either during direct monitoring or using audio recording of 1 randomly chosen session per patient or up to 8 sessions per counselor. Covering at least 75% of checklist items during each session is considered fidelity to the intervention protocol.

SECONDARY OUTCOMES:
Mental health: changes in CMD symptom response | From enrollment to the end of intervention at 6 weeks
  The mental health outcome is defined to be common mental disorders symptom response and measured as a composite score. Common mental disorders symptom response is based on common mental disorders symptom improvement. Common mental disorders symptom improvement is defined as the percent improvement in each depression, anxiety and stress subscale of the 21-item Depression, Anxiety and Stress Scale (DASS-21) from baseline, averaged across only those subscales that were elevated at baseline. Each subscale ranges from 0 to 42, with higher scores indicating worse outcomes.
Meth use: self-reported changes in meth use behaviors | From enrollment to the end of intervention at 6 weeks
  Meth use outcomes include changes in the Alcohol, Smoking and Substance Involvement Screening Test (ASSIST) score for meth and the amphetamine use behaviors scale between baseline and follow-up visits. The ASSIST score ranges from 0 to 39 for each drug assessed, higher scores indicating greater risk.
Meth use: changes in urinalysis | From enrollment to the end of intervention at 6 weeks
  Changes in the number of participants with positive urinalysis between baseline and follow-up visits.

CONTACTS AND LOCATIONS:
Locations (1):
- Friendship Bench & Lighthouse, Haiphong, Hai Phong, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tran HV, Nong HTT, Tran TTT, Filipowicz TR, Landrum KR, Pence BW, Le GM, Nguyen MX, Chibanda D, Verhey R, Go VF, Ho HT, Gaynes BN. Adaptation of a Problem-solving Program (Friendship Bench) to Treat Common Mental Disorders Among People Living With HIV and AIDS and on Methadone Maintenance Treatment in Vietnam: Formative Study. JMIR Form Res. 2022 Jul 8;6(7):e37211. doi: 10.2196/37211. PMID 35802402
- [Background] Chibanda D, Weiss HA, Verhey R, Simms V, Munjoma R, Rusakaniko S, Chingono A, Munetsi E, Bere T, Manda E, Abas M, Araya R. Effect of a Primary Care-Based Psychological Intervention on Symptoms of Common Mental Disorders in Zimbabwe: A Randomized Clinical Trial. JAMA. 2016 Dec 27;316(24):2618-2626. doi: 10.1001/jama.2016.19102. PMID 28027368
- [Background] Chibanda D. Reducing the treatment gap for mental, neurological and substance use disorders in Africa: lessons from the Friendship Bench in Zimbabwe. Epidemiol Psychiatr Sci. 2017 Aug;26(4):342-347. doi: 10.1017/S2045796016001128. Epub 2017 Apr 12. PMID 28399952
- [Background] Chibanda D, Mesu P, Kajawu L, Cowan F, Araya R, Abas MA. Problem-solving therapy for depression and common mental disorders in Zimbabwe: piloting a task-shifting primary mental health care intervention in a population with a high prevalence of people living with HIV. BMC Public Health. 2011 Oct 26;11:828. doi: 10.1186/1471-2458-11-828. PMID 22029430
- [Background] Giang HT, Duc NQ, Khue PM, Quillet C, Oanh KTH, Thanh NTT, Vallo R, Feelemyer J, Vinh VH, Rapoud D, Michel L, Laureillard D, Moles JP, Jarlais DD, Nagot N, Huong DT. Gender Differences in HIV, HCV risk and Prevention Needs Among People who Inject drug in Vietnam. AIDS Behav. 2023 Jun;27(6):1989-1997. doi: 10.1007/s10461-022-03932-x. Epub 2022 Nov 28. PMID 36441408
- [Background] Michel L, Des Jarlais DC, Duong Thi H, Khuat Thi Hai O, Pham Minh K, Peries M, Vallo R, Nham Thi Tuyet T, Hoang Thi G, Le Sao M, Feelemyer J, Vu Hai V, Moles JP, Laureillard D, Nagot N; DRIVE Study Team. Intravenous heroin use in Haiphong, Vietnam: Need for comprehensive care including methamphetamine use-related interventions. Drug Alcohol Depend. 2017 Oct 1;179:198-204. doi: 10.1016/j.drugalcdep.2017.07.004. Epub 2017 Aug 2. PMID 28800503
- [Background] Kittirattanapaiboon P, Srikosai S, Wittayanookulluk A. Methamphetamine use and dependence in vulnerable female populations. Curr Opin Psychiatry. 2017 Jul;30(4):247-252. doi: 10.1097/YCO.0000000000000335. PMID 28426546
- [Background] Tracy D, Hahn JA, Fuller Lewis C, Evans J, Briceno A, Morris MD, Lum PJ, Page K. Higher risk of incident hepatitis C virus among young women who inject drugs compared with young men in association with sexual relationships: a prospective analysis from the UFO Study cohort. BMJ Open. 2014 May 29;4(5):e004988. doi: 10.1136/bmjopen-2014-004988. PMID 24875490
- [Background] Des Jarlais DC, Feelemyer JP, Modi SN, Arasteh K, Hagan H. Are females who inject drugs at higher risk for HIV infection than males who inject drugs: an international systematic review of high seroprevalence areas. Drug Alcohol Depend. 2012 Jul 1;124(1-2):95-107. doi: 10.1016/j.drugalcdep.2011.12.020. Epub 2012 Jan 17. PMID 22257753
- [Background] Azim T, Bontell I, Strathdee SA. Women, drugs and HIV. Int J Drug Policy. 2015 Feb;26 Suppl 1(0 1):S16-21. doi: 10.1016/j.drugpo.2014.09.003. Epub 2014 Sep 17. PMID 25277726